CLINICAL TRIAL: NCT06701955
Title: Study of the Test-retest Reliability of the Neuropsychiatric Fluctuations Scale (EFN)
Brief Title: Study of the Test-retest Reliability of the Neuropsychiatric Fluctuations Scale in Parkinson's Disease
Acronym: EFN-RETEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 38RC24.0196; 2024-A01403-44 (Other: ID RCB)
Record Dates: First submitted 2024-11-19; First posted 2024-11-22 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Parkinson's Disease
Keywords: neuropsychiatric fluctuations; scale validation; psychometric caracteristics; non-motor symptoms
MeSH Terms: interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sequence of intervention (Other): self administered questionnaires at different time points..
  Interventions: Other: Questionnaire and Physical Exam

INTERVENTIONS:
Other: Questionnaire and Physical Exam — self administered questionnaires

SUMMARY:
This study focuses on neuropsychiatric fluctuations (NPF) in Parkinson's disease. Due to the lack of specific assessment tools, we developed the Neuropsychological Fluctuations Scale (NFS), a 20-item questionnaire. Recent studies have confirmed its reliability, sensitivity, and validity. To finalize its validation, assessing its test-retest reliability is an essential next step.

DETAILED DESCRIPTION:
During the progression of Parkinson's disease, a large number of patients experience fluctuations in motor status associated with neuropsychiatric fluctuations (NPF) (alternating episodes of depression, anxiety, and apathy with hypomanic states, impulsivity, and attention disorders). NPF may have a significant impact on patients' quality of life as well as on that of their caregivers. Moreover, the presence of these fluctuations is a risk factor for the development of self-medication behaviors, which can lead to addiction to antiparkinsonian treatments.

Due to the lack of specific tools for assessing NPF, our team developed a 20-item self-questionnaire specifically evaluating NPF in acute phases: the Neuropsychological Fluctuations Scale (NFS), which was first published in Movement Disorders, Clinical Practice (Schmitt et al., 2018). Recently, we studied the psychometric properties of the NFS in two populations of Parkinson's disease patients and in the general population (EFN Pre-Validation and EFN-Validation studies: ClinicalTrials.gov NCT04455074). The results regarding internal consistency, sensitivity, and specificity of the NFS, as well as its internal structure and external validity, were published in Frontiers in Neurology in 2023 (Schmitt et al., 2023). It has been demonstrated that the NFS is an innovative tool that complements existing motor and non-motor evaluations, and its utility in diagnosing and managing NPF is significant.

In order to finalize the validation of the NFS and further understand its psychometric characteristics, assessing the temporal stability of the NFS through test-retest reliability is an essential step.

ELIGIBILITY:
Inclusion Criteria:

Age > 30 and ≤ 75 years

* Idiopathic Parkinson's disease (according to the criteria of the Movement Disorders Society)
* Presence of motor fluctuations described by the patient, their relatives, or identified by the clinician
* Stability of antiparkinsonian treatment for at least one month
* Mastery of the French language
* Able to give consent.
* Affiliated to the social security system

Exclusion Criteria:

Parkinsonian syndrome other than idiopathic Parkinson's disease

* Dementia (MoCa < 23)
* No antiparkinsonian treatment or treatment modified for less than one month
* Persons referred to in Articles L1121-5 to L1121-8 of the CSP (corresponds to all protected persons: pregnant women, parturients, breastfeeding mothers, persons deprived of liberty by judicial or administrative decision, persons receiving psychiatric care under Articles L. 3212-1 and L. 3213-1 who are not covered by the provisions of Article L. 1121-8, persons admitted to a health or social establishment for purposes other than research, minors, persons subject to a legal protection measure or unable to express their consent))
* Subject in a period of exclusion from another interventional study.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
validation of test-retest reliabililty | 4 weeks
  validation of test-retest reliabililty of the neuropsychiatric fluctuations scale

CONTACTS AND LOCATIONS:
Locations (1):
- CHUGA, Grenoble, France

IPD SHARING:
Plan to Share IPD: No